CLINICAL TRIAL: NCT04530721
Title: Investigation of Multiple Ultrasound Techniques for the Assessment of Carotid Plaque Vulnerability
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-460
Record Dates: First submitted 2020-06-26; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-06

CONDITIONS: Arteriosclerosis
Keywords: ultrasound
MeSH Terms: conditions — Arteriosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stroke group
  Interventions: Other: no intervention
- normal group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — we don't do any intervention

SUMMARY:
Stroke is a common clinical disease with high disability and mortality, which seriously threatens human life and health.Carotid atherosclerotic plaque rupture is an important pathogenic basis of ischemic stroke, so judging the stability of plaque has important clinical significance in preventing ischemic stroke.Ultrasound, as a convenient, rapid, noninvasive, radiation-free auxiliary examination technology, is widely used in carotid plaque stability examination.At present, there are many methods to judge the stability of carotid plaque based on ultrasound, including two-dimensional ultrasound, contrast-enhanced ultrasound, ultrasound elastography and so on. However, the results of plaque stability judgment by various technologies deviate greatly, which is not conducive to the development of standardized diagnosis and treatment strategies by clinicians.Studies have shown that because the neovascular epidermal cells in atherosclerotic plaques are imperfect, they are easy to rupture after stress, and the ruptured neovasculature will lead to intraplaque hemorrhage, thus causing plaque shedding, and eventually obstructing the cerebrovascular cause stroke.Contrast-enhanced ultrasound can sensitively detect the distribution and course of blood vessels.The plaque's softness and hardness determine its stability, while the difference of lipids, fibers and calcium in the plaque determines its softness and hardness.Real-time ultrasound elastography can provide tissue mechanical parameters, express the soft and hard of tissue with strain value, and provide important reference information for judging plaque stability.At present, elastography technology is used to reflect the hardness of plaque, so as to further judge its stability.However, the elastography parameters are prone to deviations due to the influence of the selected section and the selected region of interest.It can be seen from the above that there is currently a multi-modality method to evaluate the stability of carotid plaque using ultrasound, but there is a lack of a unified and objective reference standard for plaque stability assessment.The purpose of this study is to explore the comprehensive utilization of these modalities under the premise of optimizing each ultrasound modality to provide a unified and objective criterion for judging the stability of carotid plaque.

ELIGIBILITY:
Inclusion Criteria:

* At least one examination suggested the presence of carotid plaque
* Suitable for CEUS examination
* Voluntary enrollment in this study and signing of informed consent

Exclusion Criteria:

* Among ischemic brain rates caused by non-carotid plaque shedding
* Follow-up Lost
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient and inpatient patients with carotid plaque in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of carotid plaque stability assessment criteria based on ultrasound multimodality Technology | 2 years
  Conventional ultrasound，CEUS，

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhang, Master, Principal Investigator — Ultrasound Department; Guoqiang Mo, Master, Study Director — Ultrasound Department
Locations (1):
- Second Affiliated Hospital,School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided